CLINICAL TRIAL: NCT00115505
Title: Quality of Life, Employment and Informal Care Cost Analysis in Women Receiving Adjuvant Chemotherapy for Breast Cancer With 0-3 Positive Axillary Lymph Nodes
Brief Title: Quality of Life, Employment, and Informal Care Costs in Women Who Are Receiving Chemotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-70301; CALGB-70301; NCI-2015-00210 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA031946 (NIH); CDR0000433266 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Breast Carcinoma
Keywords: stage IA breast cancer; stage II breast cancer; stage IB breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (QOL, employment, informal care cost): Patients complete the QOL Assessments comprising the Subjective Significance Questionnaire, MOS Social Support Survey, Patient Preferences, CALGB Background Information, and EQ-5D and QOL Assessment Form; Employment and Informal Care Cost Assessments; and Peripheral Neuropathy of the FACT-NTX subscale at baseline, 29-42 and 57-70 days, and at 9 and 18 months. Patients meeting the cut-off score for peripheral neuropathy on the FACT-NTX subscale at 18 months complete the Symptoms in Relation to Patient Functioning Survey, FACT-NTX subscale, the EORTC QLQ-C30, EORTC QLQ-BR23, and the Medications Used for Treating Peripheral Neuropathy at 24, 36, 48, and 60 months.
  Interventions: Other: quality-of-life assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: quality-of-life assessment — Complete Subjective Significance Questionnaire, MOS Social Support Survey, Patient Preferences, CALGB Background Information, and EQ-5D and QOL Assessment Form, EORTC QLQ-C30 and EORTC QLQ-BR23
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete the Employment and Informal Care Cost Assessment and Peripheral Neuropathy Assessments

SUMMARY:
This research trial studies quality of life, employment, and informal care cost analysis in patients with breast cancer receiving chemotherapy. This trial assesses how quality of life has been affected by cancer, if cancer and its treatment have caused in changes in the patient's or their spouse's employment and how they have affected the patient and their extended family, and the impact of peripheral neuropathy caused by chemotherapy on quality of life. Learning about quality of life and informal care costs may help doctors better understand how patients feel during treatment, what effects the medicines are having, and in the future may help both patients and doctors as they decide which medicines to use to treat cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the individual treatment arms relative to the degree that symptoms interfere with patient functioning and to characterize and compare the relative duration that symptoms interfere with patient functioning.

II. To assess the employment consequences of cancer and its treatment on the patient and extended family, and to compare treatment arms relative to these consequences.

III. To determine the prevalence and severity of peripheral neuropathy in breast cancer patients treated by adjuvant chemotherapy with dose dense (every two weeks) paclitaxel for 4 cycles, from study entry to 5 years after the start of treatment.

SECONDARY OBJECTIVES:

I. To identify baseline characteristics that are predictive for patients being more vulnerable to experiencing side effects which significantly interfere with patient functioning.

II. To identify and characterize the relative importance of the reasons that patients decide to participate in the treatment study (Cancer and Leukemia Group B [CALGB] 40101) and how those reasons might change as a consequence of their experience with treatment.

III. To compare the quality-adjusted life years between adjuvant chemotherapy (AC) and paclitaxel or between short and long schedules, regardless of the other factor.

IV. To measure, over the course of adjuvant therapy, the type and amount of informal care needs of the patient.

V. Using a societal perspective, estimate and compare the economic consequences on employment and informal care needs.

VI. To determine if specific identifiable clinical adverse events (i.e., neuropathy or fatigue) are associated with greater economic consequences.

VII. To examine factors which are predictive of a patient being employed during and after cancer treatment.

VIII. To compare the prevalence and severity of peripheral neuropathy in breast cancer patients treated by dose dense paclitaxel to those patients treated with dose dense CA (cyclophosphamide and doxorubicin).

IX. To conduct an exploratory examination of the relationship between the severity of peripheral neuropathy after paclitaxel treatment (4 and 6 cycles) and breast cancer patients' functioning, including physical, psychological, and social functioning.

X. To validate the neurotoxicity items in the Symptoms in Relation to Patient Functioning Survey (C-1271) used in this protocol by correlating its results with the Functional Assessment of Cancer Therapy (FACT)-Neurotoxicity Subscale (C-669) and the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core (C)30 and Breast Cancer module (C-259 and C-618).

OUTLINE:

Patients complete the QOL Assessments comprising the Subjective Significance Questionnaire, Medical Outcome Study (MOS) Social Support Survey, Patient Preferences, CALGB Background Information, and European Quality of Life 5-Dimensions (EQ-5D) and QOL Assessment Form; Employment and Informal Care Cost Assessments; and Peripheral Neuropathy of the FACT-NTX subscale at baseline, 29-42 and 57-70 days, and at 9 and 18 months. Patients meeting the cut-off score for peripheral neuropathy on the FACT-NTX subscale at 18 months complete the Symptoms in Relation to Patient Functioning Survey, FACT-NTX subscale, the EORTC QLQ-C30, EORTC QLQ-BR23, and the Medications Used for Treating Peripheral Neuropathy at 24, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be registered to CALGB 40101
* Patient must be able to communicate in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer with 0-3 positive axillary lymph nodes receiving adjuvant
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2005-10; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Degree that symptoms interfere with patient functioning according to the National Cancer Institute (NCI) Common Toxicity Criteria | Up to 18 months
Relative duration that symptoms interfere with patient functioning according to the NCI Common Toxicity Criteria | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Bunnell, MD, Study Chair — Dana-Farber Cancer Institute
Locations (227):
- United States (227):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Memorial Medical Center, Modesto, California
  - Mercy Regional Cancer Center at Mercy Medical Center, Redding, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee, Kansas
  - Cancer Resource Center at King's Daughters Medical Center, Ashland, Kentucky
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Nashville Oncology Associates, PC, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming